CLINICAL TRIAL: NCT03433612
Title: A Novel Method of Improving Accuracy of Anatomical Landmarks for Neuraxial Blocks in Pregnancy: The Sacral Anatomical Interspace Landmark (SAIL) Technique
Brief Title: Improving Accuracy of Landmarks for Neuraxial Blocks in Pregnancy: The Sacral Anatomical Interspace Landmark (SAIL) Technique
Acronym: SAIL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Carlo Pancaro, Director of Obstetrical Anesthesiology, University of Michigan
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: HUM00109509
Record Dates: First submitted 2018-02-08; First posted 2018-02-14 (Actual); Last update posted 2018-11-01 (Actual); Status verified 2018-10

CONDITIONS: Pregnancy Related
Keywords: Anatomical Landmarks
MeSH Terms: interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: All patients will undergo estimation of the L4-L5 interspace using the classic and novel technique, followed by identification of the interspace using lumbar ultrasound.
Masking Description: The estimation marks from each technique (two total) will be on the back of the patient (one on the left flank, one on the right flank), therefore the patient does not know where the marks are. Additionally, each mark will be covered with a taped on gauze pad to conceal it so that the two investigators are blinded to each others assessment. The ultrasound clinician will be masked to the two estimations. The marks will still remain covered while the interspace is determined by the third assessor using lumbar ultrasound.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- All Patients (Other): Estimates of the location of the L4-L5 intervertebral space will be done by the classic intercristal line technique and novel SAIL technique. Each technique will be performed by different randomly assigned investigators.
  * Both techiques will be assessed on all patients
  Interventions: Other: Classic Intercristal Line Technique; Other: Novel SAIL Technique

INTERVENTIONS:
Other: Classic Intercristal Line Technique — Researcher will use the classic technique to estimate the L4-L5 interspace. The classic technique begins by palpating both the right and left posterior iliac crests and following the imaginary line that intersects each (intercristal line) with the non-dominant hand to the spine where it is estimated to intersect the L4 spinous process or L4-L5 interspace. A marker pen will mark an "X" lateral to the estimation, opposite side from the estimation of the other technique.
  Other Names: Standard of Care
Other: Novel SAIL Technique — Researcher will use the novel technique to estimate the L4-L5 interspace. The SAIL technique begins by palpating the sacrum and the researcher sliding the non-dominant hand up the dorsal surface of the sacrum to the first interspace (L5-S1) and then up one more interspace to estimate the L4-L5 interspace. A marker pen will mark an "X" lateral to the estimation, opposite side from the estimation of the other technique.
  Other Names: Experimental

SUMMARY:
This study is a randomized clinical trial to evaluate the accuracy of the novel SAIL technique compared to the classic intercristal line technique in estimating the L4-L5 interspace for labor epidural or spinal anesthesia placement. The investigators hypothesize that the SAIL technique will be more accurate in successfully locating the L4-L5 interspace in pregnant women than the classic intercristal line technique.

DETAILED DESCRIPTION:
The current standard technique aiming at identifying the L4-L5 intervertebral space as a reference point before performing a neuraxial block relies on the correct clinical estimation of the intercristal line. The classic intercristal line technique uses an imaginary line that intersects the iliac crests to determine a safe puncture level to access. In pregnant women, the classic technique fails to identify the safe puncture level 40 % of the time.

The newly proposed Sacral Anatomical Interspace Landmark (SAIL) technique consists of using the sacral bone to determine a safe puncture level to access.

Lumbar ultrasound will determine the accuracy of each clinical technique in identifying the L4-L5 interspace (target).

ELIGIBILITY:
Inclusion Criteria:

* Ultrasound-determined gestation age greater than or equal to 37 weeks
* Expressed interest or indication for epidural anesthesia
* Patients in the first stage of labor

Exclusion Criteria:

* Patients perceived or indicating that she is unable to cooperate with positioning
* BMI greater than 45 kg/m2
* Previous spine surgery or known spinal deformities
* Impaired decision making abilities
* non-English speaking

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2018-02-15 (Actual); Primary Completion 2018-06-28 (Actual); Study Completion 2018-10-30 (Actual)

PRIMARY OUTCOMES:
Accuracy, as measured by percentage of estimations that correctly match ultrasound determined interspace | From enrollment to the end of data collection, approximately 15 minutes
  Percentage of trials for the novel and classic technique respectively that the estimation correctly matches the L4-L5 interspace as determined by lumbar paramedian ultrasound will serve as a measure of accuracy

CONTACTS AND LOCATIONS:
Overall Officials: Carlo Pancaro, MD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pancaro C, Rajala B, Vahabzadeh C, Cassidy R, Klumpner TT, Kountanis JA, McCabe M, Rector D, Aman C, Sankar K, Schoenfeld R, Engoren M. Sacral anatomical interspace landmark for lumbar puncture in pregnancy: A randomized trial. Neurology. 2020 Feb 11;94(6):e626-e634. doi: 10.1212/WNL.0000000000008749. Epub 2019 Dec 12. PMID 31831599